CLINICAL TRIAL: NCT07206979
Title: An Open Label Trial Assessing the Impact of a Hydration Formula on Overall Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX_OL_2505_LIV
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hydration

STUDY DESIGN:
Intervention Model Description: Eligible participants completing pretest/baseline will be stratified based on their sex assignment at birth and age then randomized to one of the study groups sequentially based on all stratification measures collectively to ensure equal distribution to each study product group. Participants will be provided the study product and the study insert with instructions for use and study participation.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Product 1 (Experimental): Hydration Active Product 1
  Interventions: Dietary Supplement: Hydration Active Product 1
- Active Product 2 (Experimental): Hydration Active Product 2
  Interventions: Dietary Supplement: Hydration Active Product 2
- Active Product 3 (Experimental): Hydration Active Product 3
  Interventions: Dietary Supplement: Hydration Active Product 3

INTERVENTIONS:
Dietary Supplement: Hydration Active Product 1 — Participants will use their Hydration Active Product 1 as directed for a period of 1 week.
  Arms: Active Product 1
Dietary Supplement: Hydration Active Product 2 — Participants will use their Hydration Active Product 2 as directed for a period of 1 week.
  Arms: Active Product 2
Dietary Supplement: Hydration Active Product 3 — Participants will use their Hydration Active Product 3 as directed for a period of 1 week.
  Arms: Active Product 3

SUMMARY:
An Open Label Trial Assessing the Impact of a Hydration Formula on Overall Health

DETAILED DESCRIPTION:
This is an open label study conducted with adult participants residing in the United States.

Eligible participants will (1) agree to consume a hydration product, (2) agree not to take any other hydration or electrolyte supplements for the duration of the trial, (3) be 21 years of age or older, and (4) agree to participate in this study for 2 week and answer assessments.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants over 2 weeks. Participant reports of health indicators will be collected at screening and throughout the active period of study product use. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
3.1 Inclusion

Participants must meet all the following criteria:

* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races.
* Resides in the United States.

3.2 Exclusion

Individuals who report any of the following during screening will be excluded from participation:

* Report being pregnant, trying to become pregnant, or breastfeeding.
* Unable to provide a valid US shipping address and mobile phone number
* Unable to read and understand English.
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

  * NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure.
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.

  * Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products.
* Reports the current use of electrolyte and/or hydration supplements that may limit the effects of the study products.
* Lack of reliable daily access to the internet.

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Hydration: Differences in self-reported perceptions of hydration | 2 weeks
  Hydration; Differences in self-reported perceptions of hydration as assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater feelings of hydration)

SECONDARY OUTCOMES:
Energy: Differences in self-reported perceptions of energy | 2 weeks
  Energy; Differences in self-reported perceptions of energy as assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater feelings of energy).
Jitters: Differences in self-reported perceptions of jitters | 2 weeks
  Jitters; Differences in self-reported perceptions of jitters as assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater feelings of jitters)
Focus; Differences in self-reported perceptions of focus | 2 weeks
  Focus; Differences in self-reported perceptions of focus as assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater feelings of focus)
Productivity: Differences in self-reported perceptions of productivity | 2 weeks
  Productivity; Differences in self-reported perceptions of productivity as assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater feelings of productivity)
Confidence: Differences in self-reported perceptions of confidence | 2 weeks
  Confidence; Differences in self-reported perceptions of confidence as assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater feelings of confidence).
Interest in Socializing: Differences in self-reported perceptions of socialization | 2 weeks
  Interest in Socializing; Differences in self-reported perceptions of socialization as assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater feelings of socialization)
Feeling Rested: Differences in self-reported perceptions of restfulness | 2 weeks
  Feeling Rested; Differences in self-reported perceptions of restfulness as assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater feelings of being rested)
Quality of Sleep: Differences in self-reported perceptions of sleep quality | 2 weeks
  Quality of Sleep; Differences in self-reported perceptions of sleep quality assessed by an item assessing perceptions of hydration (scale 1-5; where higher scores correspond to greater quality of sleep)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science Inc., Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — https://www.radiclescience.com